CLINICAL TRIAL: NCT01806974
Title: Multicenter, Prospective Study, on the Consequences of Anti-interleukin 6 Immunotherapy Treatment for Rheumatoid Arthritis on: - Healthy and Pathological Periodontium - The Level of Expression of Some Markers of Inflammation and Periodontal Pathogenic Bacteria in Periodontal Sulci and Periodontal Pockets
Brief Title: Consequences of Anti-interleukin 6 Immunotherapy Treatment for Rheumatoid Arthritis on Periodontium
Acronym: ParoPAR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: as the recruitment rate was very low, a futility study was conducted and it was decided to discontinue inclusions
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC12_0172
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Rheumatoid Arthritis; Periodontitis
Keywords: Periodontitis; rheumatoid arthritis; anti-interleukin 6; immunotherapy; inflammation; bacteria; periodontal sulci; periodontal pockets
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontitis; Inflammation; Periodontal Pocket | interventions — Diagnosis, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient with parodontitis (Other): Patient with rheumatoid arthritis and pparodontitis.
  Interventions: Other: oral exam and
- Patient without parodontitis (Other): Patient with rheumatoid arthritis but periodontally healthy
  Interventions: Other: oral exam and

INTERVENTIONS:
Other: oral exam and — The study will be conducted with patient presenting a rheumatoid arthritis and for which an anti IL6 biotherapy treatment is planned. Each patient will benefit a record oral exam that will evaluate his periodontal status and on a possible periodontitis associated. Bacterial samples and cytokine will be realized (in defined periodontal pocket or in the most affected periodontal pocket depending of the periodontal status of patients) before the IL6 biotherapy and 6 month after. A periodontal charting will be realized at the same time.

SUMMARY:
Rheumatoid arthritis and periodontitis are two inflammatory diseases that share many pathophysiological similarities as some inflammatory mediators like TNF-alpha, IL-1, Il-6, Il-17, Il-12 et Il-17, RANK-L, or OPG The most severe or progressive forms of rheumatoid arthritis require in 10-30% of cases, the use of biotherapies such as anti-TNF-alpha, anti CD-20 and anti-lL-6. All these treatments results in, among other things, an increased risk of infection, both viral and bacterial.

These new biotherapies could have an impact on periodontal status

* either by favouring sub gingival colonization of root surfaces by periodontal pathogenic bacteria and initiate periodontitis or exacerbate pre-existing periodontitis,
* or a positive modulation of the host response by inhibiting bone resorption of the alveolar process.

To date, very few studies have been conducted on this subject which is really a translational research, involving several medical specialties.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years presenting a rheumatoid arthritis and for which an anti IL6 biotherapy treatment is prescribed.
* At least 18 permanent teeth in the mouth at least 3 teeth with a healthy periodontal status
* Having expressed their written free and informed consent

Exclusion Criteria:

* Hypersensitivity to any of the following components : tocilizumab, saccharose, polysorbate 80, phosphate disodique dodécahydrate, phosphate monosodique dehydrate
* Severe or active infections
* Systemic Pathology affecting the immune system including Sjögren's syndrome
* Surgery in the previous month
* HIV positive
* Alcoholic
* Toxicoman
* Antibiotic treatment in the last 2 months
* Legally protected patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level | 6 month
  Gain or loss obtained by periodontal probing.

SECONDARY OUTCOMES:
Detection of periodontopathogenic germs | 6 month
  Detection of periodontopathogenic germs by RT - PCR - Q wich the bacterial samples will be made at the outset of the study and 6 month after the beginning of anti IL6 treatment.
Quantification of periodontopathogenic germs | 6 month
  Quantification of periodontopathogenic germs by RT - PCR - Q wich the bacterial samples will be made at the outset of the study and 6 month after the beginning of anti IL6 treatment.
Detection of inflammation markers in the gingival fluid | 6 month
  Detection and quantification of inflammation markers in the gingival fluid : IL-1, IL-6, IL-8, IL-10, IL-12, IL-15, IL-17, TGF- beta, TNF-alpha, IL-4 et IFn-gamma.
Quantification of inflammation markers in the gingival fluid | 6 month
  Quantification of inflammation markers in the gingival fluid : IL-1, IL-6, IL-8, IL-10, IL-12, IL-15, IL-17, TGF- beta, TNF-alpha, IL-4 et IFn-gamma.
Assessment of inflammation | 6 month
  Assessment of inflammation through Bleeding On Probing
Assessment of oral hygiene level | 6 month
  Assessment of oral hygiene level with plaque Index

CONTACTS AND LOCATIONS:
Overall Officials: Assem SOUEIDAN, Principal Investigator — Nantes UH
Locations (2):
- France (2):
  - Brest University Hospital, Brest
  - Nantes University Hospital, Nantes